CLINICAL TRIAL: NCT06263881
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Clinical Trial to Evaluate the Efficacy and Safety of Raphamin in Combined Treatment of Community-acquired Pneumonia
Brief Title: Clinical Trial of the Efficacy and Safety of Raphamin in Combined Treatment of Community-acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-009
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Community-acquired Pneumonia; Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raphamin (Experimental): Oral administration, without food. The tablet should be held in the mouth until complete dissolution.
  On the first day 8 tablets are administered using the following scheme: 1 tablet every 30 minutes in the first 2 hours (5 tablets in total within 2 hours), followed by three more tablets at regular intervals during the rest of the day. From day 2 onwards, 1 tablet taken 3 times daily. The treatment period is 7 days.
  Interventions: Drug: Raphamin
- Placebo (Placebo Comparator): Oral administration, without food. The tablet should be held in the mouth until complete dissolution.
  Placebo is administered according to the Raphamin regimen for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raphamin — Tablet for oral use.
  Other Names: MMH-407
  Arms: Raphamin
Drug: Placebo — Tablet for oral use.
  Arms: Placebo

SUMMARY:
Multicenter double-blind placebo-controlled randomized in parallel groups clinical trial.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, randomized in parallel-group trial.

The study enrolls male and female outpatients aged 18 to 65 years with typical symptoms of community-acquired pneumonia (CAP): axillary body temperature ≥38.00C, acute cough, shortness of breath (dyspnea), chest pain when breathing, fatigue, night sweats. Symptoms are associated with previous upper respiratory tract infection or acute bronchitis. The investigator assesses a prognosis and determines where the patient will receive treatment using the CRB-65 score which includes estimation of Confusion, Respiratory rate, Blood pressure, and Age (≥ 65 years) (min "0", max "4" points; only estimation "0" points is indication for outpatient treatment).

At the first visit (day 1), after signing the patient information sheet and informed consent form for participation in a clinical trial, the investigator collects complaints and medical history, conducts a physical examination and assessment of vital signs, and measures capillary blood oxygen saturation (SpO2), records comorbidities and concomitant therapies, collects blood samples for laboratory tests, and orders a dual-view chest X-ray or chest CT scan. If X-ray/CT shows no changes in the lungs or changes that are not typical for pneumonia, the patient is not included in the clinical trial. The investigator determines a therapeutic approach in compliance with the current standards.

At the first visit (day 1), patients are randomized to one of two treatment groups: patients in Group 1 receive Amoxicillin + Clavulanic acid (Amoxiclav) and Rafamine for 7 days; patients in Group 2 take Amoxiclav and Placebo for 7 days. All patients are provided with the drug Amoxiclav. In addition, all patients are provided with the antipyretic drug Paracetamol and a classic mercury-free thermometer to measure axillary temperature.

A second visit (3/4 days) is carried out 48-72 hours after the start of treatment to assess the effectiveness and safety of the initial course of antibiotic therapy. The investigator collects complaints, performs physical examination, and evaluates the vital signs and SpO2 level. If there is no response to initial antibiotic therapy, the decision about the therapeutic approach is made by the investigator. If hospitalization occurs, the patient ends participation in the study because he or she has reached the study endpoint.

If antibiotic therapy is effective, it is continued for 7 days. After 7 days of treatment, a third visit is carried out (day 8), at which the researcher collects the patient's complaints, conducts a physical examination and assessment of vital signs, measures SpO2 and prescribes a clinical blood test. If the patient meets the criteria for sufficiency of antibiotic therapy, the investigator stops prescribing the antibiotic.

If a positive response to the first course of antibiotic therapy is achieved, the patient continues to participate in the study. The patient is observed for 7 days. On day 15±1, the fourth visit is carried out, during which the researcher collects the patient's complaints, conducts a physical examination and assesses vital signs, measures SpO2 and prescribes a follow-up X-ray/CT scan. The patient returns the study drug and the investigator performs a compliance calculation. In total, patients are observed for 15 days.

The study uses an electronic patient diary (EPD) to record axillary temperature daily in the morning and evening. All temperature measurements during the study should be made with the same thermometer. The patient should bring the thermometer used for measurements to the health center visit. In addition, the patient should also use the EPD to record symptoms, if any, time of administration of the antipyretic dose, and any worsening of his/her condition (if applicable) to assess safety and record adverse events.

The investigator teaches the patient how to complete the diary at Visit 1. The EPD is available for completion throughout the patient's participation in the study.

An unscheduled visit may be made during the study if the patient's condition worsens or at the discretion of the investigator.

If clinical cure is not achieved by 15±1 days, the patient ends participation in the study because he or she has reached the study endpoint. The researcher determines the approach to further observation and treatment of the patient in accordance with current recommendations.

Subjects are permitted to take medications for concomitant medical conditions during the study, with the exception of medications listed in the Prohibited Concomitant Treatments section.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-65 years.
2. The diagnosis of community-acquired pneumonia presupposes that the patient has focal infiltration of the lung tissue, confirmed by imaging (X-ray/CT), and the presence of at least two clinical symptoms:

   а) acute fever at the onset of the disease (axillary temperature ≥ 38.0°C); b) wet cough; c) physical signs (crepitus/wheezing, bronchial breathing sounds, local dullness to percussion); d) leukocytosis >10×10^9/L and/or shift of band neutrophils (>10%).
3. SpO2 ≥95% according to pulse oximetry.
4. Overall CRB-65 score "0" points.
5. Patients willing to use reliable methods of contraception during the study (men and women of reproductive potential).
6. Patients who have signed the patient information sheet and informed consent.

Exclusion Criteria:

1. Any indications for patient hospitalization.
2. Suspected infiltrative pulmonary tuberculosis.
3. Medical history of/suspected malignant neoplasm of any location, including primary lung cancer and metastases to the lung parenchyma.
4. Suspected pulmonary embolism and pulmonary infarction.
5. Medical history of chronic obstructive pulmonary disease, bronchial asthma, chronic respiratory failure.
6. Medical history of immune system diseases: systemic vasculitis, lupus pneumonitis, allergic bronchopulmonary aspergillosis, obliterating bronchiolitis, idiopathic pulmonary fibrosis, eosinophilic pneumonia, bronchocentric granulomatosis.
7. Chronic heart failure III or IV FC (according to the New York Heart Association classification, 1964).
8. Suspicion of drug-induced (toxic) pneumopathy, aspiration of foreign body, sarcoidosis, pulmonary alveolar proteinosis, lipoid pneumonia, rounded atelectasis.
9. Exacerbated or decompensated chronic diseases, including diabetes mellitus, affecting a patient's ability to participate in the clinical trial.
10. Prior diagnosis of immunodeficiency of any etiology.
11. Patients having unstable angina pectoris or myocardial infarction in the previous 6 months.
12. Prior history of chronic kidney disease (categories С3-5 А3).
13. Prior history of hepatic failure (Child-Pugh class C).
14. Any surgery within the previous 3 months.
15. Patients who received any medicine specified in the section "Prohibited concomitant treatment" within 3 months preceding the inclusion in this study or who require the use of medicines that are prohibited within this trial.
16. Malabsorption syndrome, including congenital or acquired lactase deficiency (or any other disaccharidase deficiency) and galactosemia.
17. Hypersensitivity to any of the components of medications used in the treatment.
18. Pregnancy, breast-feeding; childbirth less than 3 months prior to the inclusion in the trial, unwillingness to use contraceptive methods during the trial.
19. Patients who, from the investigator's point of view, will not comply with study monitoring requirements or with study drug administration requirements.
20. Prior history of a psychiatric disorder, alcoholism or drug abuse, which in the opinion of the investigator may compromise compliance with the study protocol.
21. Participation in other clinical studies within 3 month prior to enrollment in the study.
22. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. 'Immediate relative' means husband, wife, parents, children, or siblings, regardless of whether they are natural or adopted.
23. Patients who work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e. the company's employees, temporary contract employees, persons designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with clinical cure at the test of cure (TOC) visit | On 8 days
  Percentage of patients with clinical cure at the TOC visit (on day 8 after randomization based on the physician's assessment of clinical symptoms).

SECONDARY OUTCOMES:
Average duration of antibacterial therapy | 15 days
  Average duration of antibacterial therapy in two groups

OTHER OUTCOMES:
Proportions of patients with a positive response to the initial course of antibiotic therapy after 48-72 hours | 3 days
  Proportion of patients with a positive response to the initial course of antibiotic therapy after 48-72 hours in two groups.
  The main criteria for the effectiveness of the starting regimen of antibacterial therapy after 48-72 hours: a decrease in temperature (below 38.0C), a decrease in the severity of intoxication syndrome and the main clinical symptoms of pneumonia, primarily shortness of breath.
Proportion of patients who discontinue antibiotic therapy after 7 days of treatment (based on physician assessment of clinical symptoms). | 7 days
  Proportions of patients who discontinue antibiotic therapy after 7 days of treatment in two groups (based on physician assessment of clinical symptoms).
  Criteria for the sufficiency of antibacterial therapy (all of the following must be present):
  * persistent decrease in body temperature ≤37.2ºС for at least 48 hours;
  * absence of intoxication syndrome;
  * respiratory rate <20/min (in patients without chronic respiratory failure);
  * absence of purulent sputum (except for patients with its constant secretion);
  * the number of leukocytes in the blood <10×109/l, neutrophils <80%, young forms <6%.
Proportion of patients who required a change in antibiotic 48-72 hours after initiation of therapy. | 3 days
  Proportions of patients who required a change in antibiotic 48-72 hours after initiation of therapy in two groups due to treatment failure.
  The main criteria for the treatment failure: temperature higher than 38.0C), presence of intoxication syndrome and the main clinical symptoms of pneumonia, shortness of breath.
Time until a persistent decrease in body temperature ≤37.2ºС (according to the patient's diary). | 15 days
  Time until a persistent decrease in body temperature ≤37.2ºС (according to the patient's diary) in two groups.
Proportion of patients who required a second course of antibiotic therapy. | 15 days
  Proportions of patients who required a second course of antibiotic therapy in two groups due to treatment failure.
  The main criteria for the treatment failure: temperature higher than 38.0C), presence of intoxication syndrome and the main clinical symptoms of pneumonia, shortness of breath.
Proportion of patients who required hospitalization during 15 days of follow-up. | 15 days
  Proportions of patients who required hospitalization during 15 days of follow-up due to treatment failure.
  The main criteria for the treatment failure: temperature higher than 38.0C), presence of intoxication syndrome and the main clinical symptoms of pneumonia, shortness of breath.
Number of antipyretic drug doses taken during 7 days of the initial course of antibacterial therapy (per patient). | 7 days
  Average number of antipyretic drug doses taken during 7 days of the initial course of antibacterial therapy (per patient) in two groups according to the patient's diary.
Proportion of patients without infiltration on x-ray/CT 14 days after randomization. | 14 days
  Proportions of patients without infiltration on X-ray/CT on 14th day after randomization in two groups according to medical records.
The Presence of Adverse Events (AEs). | 15 days
  The presence and nature of adverse events, their intensity (severity), causal relationship to the study drug, outcome. Based on medical records.
Changes in Vital Signs (Blood Pressure measured in mm Hg) | 15 days
  Changes in Blood Pressure at the end of treatment. Based on medical records.
Changes in Vital Signs (Pulse Rate (Heart Rate) measured in beats per minute) | 15 days
  Changes in Heart Rate at the end of treatment. Based on medical records.
Changes in Vital Signs (Respiratory Rate (Breathing Rate) measured in breaths per minute) | 15 days
  Changes in Respiratory Rate at the end of treatment. Based on medical records.

CONTACTS AND LOCATIONS:
Locations (38):
- Russia (38):
  - Aramil city hospital, Aramil
  - Northern Medical Clinical Center named after N.A. Semashko Federal Medical and Biological Agency, Arkhangelsk
  - Gatchina Clinical Interdistrict Hospital, Gatchina
  - Ivanovo Clinical Hospital named after Kuvayevs, Ivanovo
  - City Clinical Hospital # 9 of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Central City Clinical Hospital, Kaliningrad
  - Kazan State Medical University/Department of Infectious Diseases, Kazan'
  - Kazan State Medical University, Kazan'
  - Kuban State Medical University/Department of Infectious Diseases and Phthisiopulmonology, Krasnodar
  - Central Research Institute of Epidemiology, Moscow
  - First Moscow State Medical University named after I.M. Sechenov, Moscow
  - Moscow Regional Research Clinical Institute named after. M.F. Vladimirsky, Moscow
  - Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko, Nizhny Novgorod
  - LLC "Persona group of companies", Nizhny Novgorod
  - Clinical Hospital # 4, Penza
  - LLC "Professor's clinic", Perm
  - Nikolaevskaya hospital, Petergof
  - LLC "4D Ultrasound Clinic", Pyatigorsk
  - Rostov Central District Hospital, Rostov
  - St. Petersburg Research Institute of Phthisiopulmonology, Saint Petersburg
  - LLC "Energy of Health", Saint Petersburg
  - LLC "Medical center "Reavita Med SPb", Saint Petersburg
  - LLC "Medical Clinic", Saint Petersburg
  - City Polyclinic # 112, Saint Petersburg
  - LLC "Zvezdnaya Clinic", Saint Petersburg
  - City Pokrovskaya Hospital, Saint Petersburg
  - City Polyclinic # 4, Saint Petersburg
  - LLC "Meili", Saint Petersburg
  - Medical University "Reaviz", Samara
  - Samara State Medical University/Department of General and Clinical Microbiology, Immunology and Allergology, Samara
  - Smolensk State Medical University, Smolensk
  - LLC "Scientific Medical Center of General Therapy and Pharmacology", Stavropol
  - Bashkir State Medical University/Department of Internal Medicine, Ufa
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Regional Clinic Hospital, Vladimir
  - Voronezh Regional Clinical Hospital # 1, Voronezh
  - Clinical Hospital # 2, Yaroslavl
  - LLC "Medical Center for Diagnostics and Prevention Plus", Yaroslavl

IPD SHARING:
Plan to Share IPD: No